CLINICAL TRIAL: NCT04888026
Title: Impact on Pain Sensitivity of Clinical Interaction
Acronym: QSTROBOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spine Centre of Southern Denmark (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: QSTROBOT
Record Dates: First submitted 2021-03-22; First posted 2021-05-17 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Pain Measurement
Keywords: Low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Automated QST procedure (Experimental): The QST robot will autonomously perform i) pressure pain thresholds at the tibialis anterior, ii) the cold-pressor test, and iii) repeat the pressure pain threshold. All verbal information is giving through the computer
  Interventions: Device: Quantitative sensory testing
- Manual QST procedure (Active Comparator): The research assistant will perform i) pressure pain thresholds at the tibialis anterior, ii) the cold-pressor test, and iii) repeat the pressure pain threshold. All tests are performed manually without using the robot.
  Interventions: Device: Quantitative sensory testing
- Semi-automated QST procedure (Active Comparator): The QST robot will with guidance from the research assistant perform i) pressure pain thresholds at the tibialis anterior, ii) the cold-pressor test, and iii) repeat the pressure pain threshold. However and in contrast to the first arm, all verbal information and procedure guiding is given by a research assistant.
  Interventions: Device: Quantitative sensory testing

INTERVENTIONS:
Device: Quantitative sensory testing — The following QSTs are conducted:
  The pressure pain threshold on the tibialis anterior
  The Cold-pressor test
  Repeat of the pressure pain threshold to assess conditioned pain modulation

SUMMARY:
Pain can currently be quantified using quantitative sensory tests (QSTs). However, we lack knowledge concerning how relational and contextual factors impact these quantitative tests. We will examine how a standard QST battery is affected by "removing" the social and human interaction from the test session compared to usual QST testing where the participant is guided through the assessment by a research assistant.

Our objectives are:

1. How is the QST affected when guided by a research assistant compared to guided by a computer
2. Does the level of the assessor's empathy affect the QST outcome
3. How do psychological factors affect the QST testing
4. are these outcomes affected by the patient profile (low back pain patients vs healthy controls)

ELIGIBILITY:
Inclusion Criteria:

* Primary complaint of low back pain
* No pain for healthy controls
* No serious psychological or somatic disorders potentially interfering with the QST

Exclusion Criteria:

* Incomplete QST data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
The Conditioned pain modulation effect [changes in kPa] | Baseline
  Between-group differences in conditioned pain modulation (CPM). The CPM [range -1000;1000 kPa] is measured as the change between a pressure pain threshold test before and after a cold pressor test (2 minutes of immersion the left hand in ice water].

SECONDARY OUTCOMES:
Pressure pain threshold | Baseline
  Between-group differences in pressure pain threshold [range 0-1000 kPa] as measured before the cold pressor test

CONTACTS AND LOCATIONS:
Overall Officials: Søren Neill, PhD, Principal Investigator — Director of research
Locations (3):
- Denmark (3):
  - Spine Centre of Southern Denmark, Middelfart
  - The Spine Center of Southern Denmark, Middelfart
  - Department of Physocolgy, Odense

IPD SHARING:
Plan to Share IPD: No
Data is available upon reasonable request after the pre-planned analysis are performed

REFERENCES:
- [Derived] Nim CG, Ravn SL, Andersen TE, Engelsholm E, Hestbech F, Hvidkaer IS, Traidl AN, O'Neill S. No effect of social interaction on experimental pain sensitivity: a randomized experimental study. Pain. 2023 Sep 1;164(9):2112-2121. doi: 10.1097/j.pain.0000000000002913. Epub 2023 Apr 13. PMID 37058414